CLINICAL TRIAL: NCT05988931
Title: Comparing Scalable Technology-Driven Brief Intervention Packages for Youth Alcohol Use
Brief Title: Technology Interventions for Youth Alcohol Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Maureen A Walton, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00232130; AU-2022C1-25631 (Other: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Web Program + App (Active Comparator): Brief intervention web program (rooted in Motivational Interviewing) recommended at enrollment with parent/caregiver recommended to download and use app (with strategies to talk to youth about drinking prevention).
  Interventions: Behavioral: Web Program + App
- Web Program + App + Text Messages (Active Comparator): Brief intervention web program (rooted in Motivational Interviewing) recommended at enrollment with parent/caregiver recommended to download and use app (with strategies to talk to youth about drinking prevention) plus youth receive 8 weeks of text messages.
  Interventions: Behavioral: Web Program + App + Text Messages

INTERVENTIONS:
Behavioral: Web Program + App — Youth receive a brief interactive web program made available online to prevent alcohol misuse. The parent/caregiver app addresses monitoring and skill building for parents to communicate with the child about preventing underage drinking and drug use.
  Arms: Web Program + App
Behavioral: Web Program + App + Text Messages — Youth receive a brief interactive web program made available online to prevent alcohol misuse. This is followed by 8 weeks of supportive text messages. The parent/caregiver app addresses monitoring and skill building for parents to communicate with the child about preventing underage drinking and drug use.
  Arms: Web Program + App + Text Messages

SUMMARY:
The purpose of this study is to evaluate the effects of two programs to prevent/reduce alcohol misuse among youth primary care patients. Depending on their study condition, youth will receive a brief web-based computer program or the web program + 8 weeks of supportive text messages. Parents/caregivers of youth are encouraged to use a freely available app to guide conversations with their child about drinking. This study will have significant impact by evaluating response to these scalable interventions which can be deployed widely in clinical care settings.

ELIGIBILITY:
Inclusion Criteria:

* patients age 12-19 within the Michigan Medicine health system who had a visit within the past 2 years; and
* past 12-month alcohol use; and
* patient has a phone that can receive text messages

Exclusion Criteria:

* patients who do not understand English; or
* patients deemed unable to provide informed consent due to conditions that preclude understanding of assessment or intervention content; or
* parent/guardian consent is not obtained; or
* another child in household already enrolled in the study; or
* ongoing participation in another behavioral health research study

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Consumption | 3-, 6-, 9- and 12- months post baseline
  Alcohol consumption will be measured using total score on the 3-item Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) which includes typical quantity and frequency, and frequency of binge drinking (# of drinks modified by age based on the NIAAA Youth Guide). Higher score indicates worse outcomes.

SECONDARY OUTCOMES:
Change in Alcohol Related Consequences | 3-, 6-, 9- and 12- months post baseline
  Alcohol related consequences will be measured using total score on the brief 18-item version of the Rutgers Alcohol Problem Index (RAPI). Higher score indicates worse outcomes.
Change in Other Drug Use | 3-, 6-, 9- and 12- months post baseline
  Other drug use will be measured using scores derived from National Survey on Drug Use and Health (NSDUH) survey items for illicit (e.g., cannabis, cocaine, heroin) and prescription (i.e., in any way a doctor did not direct you to use; stimulants, sedatives, and opioids) drugs misuse. Higher scores indicate worse outcomes.
Change in Other Drug Use Consequences | 3-, 6-, 9- and 12- months post baseline
  Other drug use consequences will be measured using total score on an 18-item version of the drug-focused RAPI. Higher score indicates worse outcomes.
Change in Depression Symptoms | 3-, 6-, 9- and 12-month post baseline
  Depressive symptoms will be measured using the Patient Health Questionnaire-2 (PHQ-2). Higher scores indicate worse outcomes, with a score of ≥ 3 indicating a positive depression screen.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Walton, MPH, PhD, Principal Investigator — University of Michigan; Erin Bonar, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No